CLINICAL TRIAL: NCT05272527
Title: The Effect of the "Transition to Motherhood Program" Applied to Primipar Pregnants on the Process of Self-Assessment, Postpartum Problems, and Maternal Attachment: RCT
Brief Title: Postpartum Affects of Transition to Motherhood Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilknur Aydin Avci, Head of Nursing Department, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ODM.0.20.08/677-799-844
Record Dates: First submitted 2021-12-28; First posted 2022-03-09 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy
Keywords: Pregnancy; transition to motherhood; postpartum problems; maternal attachment

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): After the pre-tests were completed, the pregnant women were divided into experimental and control groups. Within the scope of the Transition to Motherhood Program, 5-session training and phone follow-ups were made in the first week and the fourth week postpartum to the experimental group. Post-tests were applied to the experimental group at the postpartum 1st month and 4th month.
  Interventions: Behavioral: Transition to Motherhood Program
- Control Group (No Intervention): After the pre-tests were completed, the pregnant women were divided into experimental and control groups. Pretest and postpartum 1st month and 4th month posttests were applied to the control group.

INTERVENTIONS:
Behavioral: Transition to Motherhood Program — Transition to Motherhood program includes 5 sessions. The first session covers the pregnancy process, the second session deals with the birth process, the third session deals with the postpartum period, the fourth session deals with infant care, and the fifth session deals with breast milk and breastfeeding and immunity. Trainings are online. In addition to the lecture technique, the training includes auxiliary techniques such as models, videos, case studies, training cards, and applied demonstrations. The program was completed by telephone follow-up in the first and fourth weeks postpartum.
  Arms: Intervention Group

SUMMARY:
It has been seen that primiparous pregnant women experience similar problems during the transition to motherhood, and these problems affect both their self-evaluation, physical problems in the postpartum period, and maternal attachment. It is thought that the correct and adequate care and training received from health professionals will be effective in the solution of all these interconnected situations.

The study aims to determine the effect of the "Transition to Motherhood Program (TMOP)" applied to primiparous pregnant women on self-assessment, postpartum problems, and maternal attachment.

MethoThis research method is a randomized, control group pretest-posttest experimental research. The population of the study consisted of pregnant women who were registered to two Family Health Centers between December 2019 and December 2021 and met the inclusion criteria, the sample consisted who agreed to participate in the study (experimental group: 38, control group: 38).In the study, Personal Information Form, Prenatal Self-Assessment Scale, Prenatal Attachment Scale were applied to all pregnant women in the sample group as pre-test applications. Based on Meleis' Transition Theory, the Transition to Motherhood Program was applied to the pregnant women in the experimental group. The post-test application of the research was carried out in the sixth weeks and fourth postpartum months. At the sixth week of the postpartum period, the Postpartum Self-Assessment Scale, Postpartum Physical Symptom Scale, Maternal Attachment Scale; at the fourth month of the postpartum period, the Maternal Attachment Scale was used. In data analysis, dependent sample t test, ki square, mann whitney u tests will use. Necessary permissions were obtained for the study.

DETAILED DESCRIPTION:
Pregnancy, which most women experience at least once, is defined as an active part of life in which natural and pathological processes are intertwined. Pregnancy begins with fertilization due to the union of male and female reproductive cells. The standard duration of pregnancy is accepted as an average of 280 days or 40 weeks from the last menstrual period. The period from the first moment of fertilization to the 12th week of pregnancy is considered the first trimester, and it is known that the risk of miscarriage is highest in this period. The period between 13 and 28 weeks is regarded as the second trimester, and the risk of pregnancy is decided in this trimester. The third trimester is between 29 weeks and approximately 40 weeks and ends with birth. The third trimester is considered to be the most trouble-free period of pregnancy. Although it is accepted as a normal physiological process, various problems such as nausea, back pain, bowel and bladder issues, skin changes, fatigue, headache, and prenatal anxiety can be experienced during pregnancy. For pregnant women who cannot cope with these problems, a psychologically damaging situation may occur during pregnancy and in the postpartum period. It is emphasized that having previous pregnancy and birth experience can reduce this effect, but primiparous (first pregnancy) pregnant women are more affected by these problems.

Those who have been pregnant for the first time or have given birth only once; women with no previous pregnancy and motherhood experience are defined as primiparous pregnant women. Studies have reported that primiparous women need training in fulfilling their roles and responsibilities in newborn care, and it takes longer for these mothers to take care of their babies. In a study conducted with primiparous pregnant women, About 82% of the participants experienced fear of childbirth, 75% were worried about body image, 74% experienced mood swings, 79% changed their lifestyle after conception, and 86% experienced depression, anxiety, stress. It has been stated that there are psychological problems. In another study, the causes of the issues experienced by primiparous pregnant women in this process; It was found that they felt inadequate, had difficulties in coping, and could not fully adapt to the transition to motherhood.

"The Transition to Motherhood" is one of the most significant developmental life events of women's lives. According to Meleis, the concept of being a mother expresses a new role transition from a known situation to another strange case. The transition to motherhood requires re-meaning the goals, behaviors, and responsibilities to gain new meanings. This transition requires reinterpreting goals, behaviors, and commitments to acquire new definitions. Transition to motherhood; It is affected by the importance that pregnant women ascribe to the process, their characteristics, their level of knowledge, skills, and well-being. Support from unsafe sources about pregnancy and motherhood can be challenging for a healthy transition to motherhood. Insufficient support, undesirable or harmful suggestions, unreliable and contradictory information, being forced to be stereotyped, negative attitudes from those around, care that ignores individuality are considered as complicating factors in this process. Facilitating factors in the transition to motherhood are listed as being ready for motherhood, receiving adequate social support, training and counseling services specific to personality traits, good role models, and being physically healthy. In addition, the definition of the role of motherhood, the positive contribution of social networks, easy access to resources, and support are shown as other facilitating factors. It is stated that pregnant women who cannot complete the transition to motherhood in a healthy way have more difficulty in adapting to motherhood. They experience a lot of fear about childbirth and evaluate themselves negatively. Although there is not enough information about the transition process and the answers given to the transitions, Meleis assumed that the area that needs improvement is not transitions but what nurses can do for these individuals to get healthy outputs after the transitions.

Since the self-evaluation status of the pregnant will affect her and her baby's mental health during the transition to motherhood, It is thought that it is essential to make positive interventions.

Research Questions

1. What descriptive and pregnancy-related characteristics of primiparous pregnant women participating in the study?
2. Does the application of "ANGEP" prepared according to Meleis' Transition theory to primiparous pregnant women affect their postpartum self-evaluation?
3. Does the application of "ANGEP," which is prepared according to Meleis' Transition theory, to primiparous pregnant women affect their physical problems in the postpartum period?
4. Does the application of "ANGEP" prepared according to Meleis' Transition theory to primiparous pregnant women affect maternal attachment status?

ELIGIBILITY:
Inclusion Criteria:

* Not being a multiple and risky pregnancy (healthy pregnant women were selected to understand the effectiveness of the training program),
* Being over the age of 18, under the age of 35 (this age range has been chosen since pregnancies younger than 18 and older than 35 are considered risky pregnancies),
* Being the first pregnancy (women who had no previous pregnancy experience were selected to better understand the effectiveness of the training),
* Being in the 24th week of pregnancy (pregnant women in this week have been selected to make it clear that the pregnancy is not risky),
* Being literate,
* Using a smart phone and not having internet access problems (required as the trainings will be held online),
* Not having a chronic disease,
* Not having a communication barrier and being willing to participate in the study,
* Not going to pregnant schools (this criterion has been set so that it does not affect the educational effectiveness).

Exclusion Criteria:

* Having a risky pregnancy,
* Previous pregnancy,
* More than 24 weeks of gestation,
* Presence of a chronic disease,
* Being illiterate,
* Pregnancy with assisted reproductive techniques,
* Not having a smart phone and/or having internet access problems,
* Going to maternity school or getting any training related to pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Prenatal Self-Assessment Scale-pretest | 3 month
  The Scale was developed by Lederman to evaluate the adaptation of women in the prenatal period to pregnancy and the role of motherhood. It hasa 79-item, 4-point Likert-type scale, and has 7 subscales. Subscales are "acceptance of pregnancy", "acceptance of the role of motherhood", "relationship with her own mother", "relationship with her spouse", "readiness for birth", "fear of birth", "thoughts about her own and her baby's health". Low scores indicate high compliance with pregnancy.
Prenatal Attachment Inventory-pretest | 3 month
  The Cronbach alpha coefficient of the scale, which was developed by Muller and Mercer (1993) to explain the thoughts, feelings and situations experienced by women during pregnancy, and to determine the level of attachment to the baby in the prenatal period, is 0.86 (Muller and Mercer, 1993). The validity and reliability study of the Turkish version of the PCI was performed by Yılmaz and Beji (2013), and the Cronbach alpha reliability coefficient was found to be 0.84 (Yılmaz & Beji, 2013). The scale consists of 21 items; Each item is of a four-point Likert type, with a score between 1 and 4. A minimum of 21 points and a maximum of 84 points can be obtained from the scale. The increase in the score obtained by the pregnant indicates that the level of attachment also increases. It is scored as 1: Never, 2: Sometimes, 3: Often, 4: Always. The increase in the score obtained by the pregnant indicates that the level of prenatal attachment also increases.
Postpartum Self-Assessment Scale-posttest | 6 month
  It is an 82-item, 4-point Likert-type scale developed by Lederman and Weingarten in 1981 to evaluate postpartum women's adjustment to motherhood. The scale has 7 subscales that evaluate postpartum adjustment of mothers. Subscales are "the quality of the relationship between the partners", "the partners' view of participation in baby care", "satisfaction with the birth experience", "satisfaction with the continuation of life", "confidence in coping with maternal duties", "satisfaction with motherhood and newborn care", "support of family and friends for motherhood". Low scores indicate high postpartum adjustment.
Postpartum Physical Symptom Severity Scale-posttest | 6 month
  The scale, developed to determine the prevalence and persistence of postpartum physical symptoms, is a 4-point Likert-type scale with a total of 18 items. "Perineal pain"," insomnia", "constipation", "back pain", "headache", "hemorrhoids", "joint pain", "hand numbness", "vaginal discharge and infection", "foot numbness", "vaginal bleeding"," urinary tract infection"," dizziness", "varicose veins in the legs", "urinary incontinence" occurring in the postpartum period assesses physical symptoms and their severity. The scale has no cut-off point and an increase in the score from the scale indicates that the severity of postpartum physical symptoms is high.
Maternal Attachment Scale-1st posttest | 6 month
  The scale developed by Muller (1994); It is applied to women who have babies between one and four months postpartum to determine maternal feelings and behaviors. The scale which measures maternal emotions and behaviors showing love, is a scale that can be applied to women who can read and write and understand what they read, as it is a self-administered scale. The scale consists of 26 questions with 4-point Likert type. All questions contain answers ranging from 'always' to 'never'; It is calculated as Always (a)=4, Often (b)=3, Sometimes (c)=2, and Never (d)=1 points. From the sum of the questions; The lowest score to be obtained varies between 26 and the highest score ranges from 104.

SECONDARY OUTCOMES:
Maternal Attachment Scale- 2nd posttest | 9 month
  The scale developed by Muller (1994); It is applied to women who have babies between one and four months postpartum to determine maternal feelings and behaviors. The scale which measures maternal emotions and behaviors showing love, is a scale that can be applied to women who can read and write and understand what they read, as it is a self-administered scale. The scale consists of 26 questions with 4-point Likert type. All questions contain answers ranging from 'always' to 'never'; It is calculated as Always (a)=4, Often (b)=3, Sometimes (c)=2, and Never (d)=1 points. From the sum of the questions; The lowest score to be obtained varies between 26 and the highest score ranges from 104.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur AYDIN AVCİ, Prof. Dr., Study Director — Ondokuz Mayıs University; Mustafa Kürşat ŞAHİN, Assoc Prof., Study Chair — Ondokuz Mayıs University; Oya Sevcan ORAK, Asist Prof, Study Chair — Ondokuz Mayıs University
Locations (1):
- Dilek ÇELİK EREN, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lederman RP, Lederman E, Work BA Jr, McCann DS. Relationship of psychological factors in pregnancy to progress in labor. Nurs Res. 1979 Mar-Apr;28(2):94-7. PMID 254068
- [Background] Muller ME. Development of the Prenatal Attachment Inventory. West J Nurs Res. 1993 Apr;15(2):199-211; discussion 211-5. doi: 10.1177/019394599301500205. No abstract available. PMID 8470375
- [Background] Muller ME. A questionnaire to measure mother-to-infant attachment. J Nurs Meas. 1994 Winter;2(2):129-41. PMID 7780768
- [Background] Chien LY, Tai CJ, Hwang FM, Huang CM. Postpartum physical symptoms and depressive symptomatology at 1 month and 1 year after delivery: a longitudinal questionnaire survey. Int J Nurs Stud. 2009 Sep;46(9):1201-8. doi: 10.1016/j.ijnurstu.2009.02.007. Epub 2009 Mar 10. PMID 19278680
- [Background] Perinatal parental behavior: nursing research and implications for newborn health. Birth Defects Orig Artic Ser. 1981;17(6):1-308. No abstract available. PMID 7326368
- [Derived] Celik Eren D, Aydin Avci I. The Impact of a Transition to Motherhood Program on Postpartum Outcomes of Primiparous Women: A Randomized Controlled Trial. Matern Child Health J. 2025 Nov;29(11):1610-1620. doi: 10.1007/s10995-025-04181-9. Epub 2025 Sep 25. PMID 40996490